CLINICAL TRIAL: NCT01252199
Title: A Phase II Study of Chimeric Monoclonal Antibodies to Shiga Toxins 1 (cαStx1) and 2 (cαStx2) Administered Concomitantly to Children With Shiga Toxin-Producing Bacterial (STPB) Infection and Bloody Diarrhea (SHIGATEC Trial)
Brief Title: Study of Chimeric Monoclonal Antibodies to Shiga Toxins 1 and 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thallion Pharmaceuticals (Industry)
Collaborators: LFB Biotechnologies, SAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTP_STX005/STX005EXT
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Shiga Toxin Producing Bacterial Infection
Keywords: Shigamabs; Monoclonal; Antibodies; Shiga; Toxin; E.coli; HUS; Bloody; Diarrhea
MeSH Terms: conditions — Escherichia coli Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cαStx1/cαStx2 (Experimental)
  Interventions: Drug: cαStx1/cαStx2
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cαStx1/cαStx2 — cαStx1/cαStx2 administered concomitantly at a dose of 1 mg/kg (low dose cohort) or 3 mg/kg (high dose cohort)per antibody over 1 hour + standard of care
  Arms: cαStx1/cαStx2
Drug: Placebo — Placebo administered over 1 hour + standard of care
  Arms: Control

SUMMARY:
This study is designed to evaluate the safety and efficacy of cαStx1 and cαStx2 administered concomitantly in children presenting early signs of Shiga Toxin-Producing Bacterial (STPB) Infection.

DETAILED DESCRIPTION:
Currently, there is no etiological treatment of STPB-induced HUS. Ideally, such treatment would be started in the early phase of the infection and would protect against both types of toxins and all of their variants. The chimeric anti-Shiga toxins 1 (cαStx1) and 2 (cαStx2) antibodies are intended to be administered as a single infusion and provide simultaneous protection against the two Shiga toxins (Stx1 and Stx2) by decreasing the incidence and severity of Shiga toxin-mediated clinical events including bloody diarrhea/hemorrhagic colitis and Hemolytic Uremic Syndrome (HUS) and associated sequelae.

ELIGIBILITY:
Inclusion Criteria:

1. Bloody diarrhea (by visual inspection) for no more than 36 hours prior to screening (signature of the informed consent).
2. Detection of Shiga toxin (Stx1 and/or Stx2) in stool

Exclusion Criteria:

1. Laboratory findings compatible with development of at least two out of three following criteria that define Hemolytic Uremic Syndrome (HUS):

   Hemolytic Anemia: hematocrit < 30% with evidence of hemolysis (as indicated by Lactate Dehydrogenase (LDH) above the upper limit of normal for age or the finding of schistocytes on peripheral smear); Thrombocytopenia: platelet count <150 x 103/uL; Nephropathy: serum creatinine > Upper Limit Normal (ULN) adjusted for age and gender.
2. Bloody-diarrhea suspected not to be caused by Shiga Toxin-Producing Bacteria (STPB) but by other organisms or preexisting diseases.
3. Family history of proven or suspected hereditary Hemolytic Uremic Syndrome (HUS) or thrombotic thrombocytopenic purpura (TTP).
4. History of chronic/recurrent hemolytic anemia or thrombocytopenia.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Evaluation of number and type of adverse events and serious adverse events between arms and dosage cohorts | Up to 1 year
  Evaluation of the safety and tolerability of two different intravenous dose levels of a combined cαStx1/cαStx2 preparation in separate groups of children presenting with Shiga Toxin-Producing Bacterial (STPB) infection.

SECONDARY OUTCOMES:
Efficacy: Comparison of clinical event rates (Hemolytic Uremic Syndrome, Bloody Diarrhea) and associated sequelae between arms and dosage cohorts in children presenting with Shiga Toxin-Producing Bacterial (STPB) infection. | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (11):
- Argentina (7):
  - Bahía Blanca
  - Buenos Aires
  - Córdoba
  - La Plata
  - Mendoza
  - Paraná
  - San Miguel de Tucumán
- Chile (3):
  - Concepción
  - Santiago
  - Valparaíso
- Lima, Peru

REFERENCES:
- [Derived] Imdad A, Nelson JR, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2025 Apr 25;4(4):CD012997. doi: 10.1002/14651858.CD012997.pub3. PMID 40277027
- [Derived] Imdad A, Mackoff SP, Urciuoli DM, Syed T, Tanner-Smith EE, Huang D, Gomez-Duarte OG. Interventions for preventing diarrhoea-associated haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Jul 5;7(7):CD012997. doi: 10.1002/14651858.CD012997.pub2. PMID 34219224